CLINICAL TRIAL: NCT06430047
Title: The Role of an EsoDuo® to Control Reflux Symptoms Related to the Acid; a Multicenter, Open-labeled, Phase 4 Study [RACER Study]
Brief Title: Efficacy and Safety of EsoDuo®
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B73_02GERD2107
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Gastro Esophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental)
  Interventions: Drug: EsoDuo® Tablet

INTERVENTIONS:
Drug: EsoDuo® Tablet — QD, PO

SUMMARY:
Clinical Trial to Evaluate the Effects of EsoDuo® in Controlling Reflux Symptoms Related to the Acid

DETAILED DESCRIPTION:
The Role of an EsoDuo® to Control Reflux Symptoms Related to the Acid; a Multicenter, Open-labeled, Phase 4 Study [RACER Study]

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female aged ≥ 19 years
2. Patients diagnosed with non-erosive reflux disease or mild erosive reflux disease
3. Episode of heartburn the GERD symptom(either heartburn or gastric acid reflux)

Exclusion Criteria:

1. Surgery history on stomach or esophagus
2. Barrett's esophagus (over 3cm), esophageal varices, esophageal stricture, esophageal achalasia, eosinophilic esophagitis, and primary motility disorders
3. Patients diagnosed with Grade C or Grade D according to the LA Classification system during upper gastrointestinal endoscopy
4. Patients with a history of malignancy within the past 5 years prior to the screening visit (Visit 1)
5. Patients who have taken prohibited concomitant medications within 14 days prior to the screening visit or require continuous administration of prohibited medications during the trial period.
6. Clinically significant Abnormal Lab test
7. Pregnant woman, Breastfeeding woman.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-11-25 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
The time taken to control the symptoms of GERD | 2 weeks after the clinical trial participation
  the symptoms of GERD : heartburn or acid reflux

CONTACTS AND LOCATIONS:
Overall Officials: Hwoon-Yong Jung, M.D, PhD, Principal Investigator — Asan Medical Cental of Korea
Locations (1):
- Asan Medical Center, Seoul, South Korea